CLINICAL TRIAL: NCT06213649
Title: Parasitic Ulcer Treatment Trial
Acronym: PUTT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jeremy Keenan, MD, MPH (Other)
Collaborators: Johns Hopkins University (Other); Oregon Health and Science University (Other); University of Illinois at Chicago (Other); University of California, Los Angeles (Other); University of Pittsburgh (Other); University of Pennsylvania (Other); Columbia University (Other); University of Iowa (Other); University of Florida (Other); Aravind Eye Care System (Other); Moorfields Eye Hospital NHS Foundation Trust (Other); Federal University of São Paulo (Other); National Eye Institute (NEI) (NIH); University of Miami (Other)
Responsible Party: Sponsor-Investigator, Jeremy Keenan, MD, MPH, Professor of Ophthalmology/Director of International Programs at the Proctor Foundation, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-39559; UG1EY033284 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Acanthamoeba Keratitis
Keywords: corneal ulcer; steroids
MeSH Terms: conditions — Acanthamoeba Keratitis; Corneal Ulcer | interventions — polihexanide; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical steroids (Experimental): Participants in this arm will receive anti-amoebic therapy plus topical steroids.
  Interventions: Drug: Polyhexamethylene biguanide (PHMB); Drug: Topical corticosteroid
- Topical placebo (Placebo Comparator): Participants in this arm will receive anti-amoebic therapy plus topical placebo.
  Interventions: Drug: Polyhexamethylene biguanide (PHMB); Other: Topical placebo

INTERVENTIONS:
Drug: Polyhexamethylene biguanide (PHMB) — PHMB is a cationic antiseptic agent used for topical treatment of acanthamoeba keratitis (AK). Both treatment groups will take PHMB at least 4 times daily while on the allocated study drug.
  Other Names: Polyhexanide
Drug: Topical corticosteroid — Dexamethasone sodium phosphate, 0.1% ophthalmic solution will be administered 4 times daily for 4 weeks, then 2 times daily for 2 weeks, then 1 time daily for 2 weeks.
  Arms: Topical steroids
Other: Topical placebo — An artificial tear ophthalmic solution will be administered 4 times daily for 4 weeks, then 2 times daily for 2 weeks, then 1 time daily for 2 weeks.
  Arms: Topical placebo

SUMMARY:
The Parasitic Ulcer Treatment Trial (PUTT) is a multi-center, parallel-group, randomized clinical trial. The purpose of this study is to determine whether including topical corticosteroids in a regimen for acanthamoeba keratitis (AK) will improve vision. Patients presenting to all enrollment centers with evidence of acanthamoeba keratitis will be eligible for the trial if there is evidence of ocular inflammation after 4 weeks of anti-amoebic therapy. Those who agree to participate will be randomized to one of two treatment groups:

* Group 1: Topical corticosteroid
* Group 2: Topical placebo

ELIGIBILITY:
Inclusion Criteria:

* AK on at least one of the following: culture, smear, PCR, shotgun sequencing, biopsy, or confocal microscopy
* Ocular inflammation after 1 month of anti-amoebic treatment, defined as conjunctival, corneal, episcleral, or anterior chamber inflammation

Exclusion Criteria:

* Evidence or history of interstitial keratitis
* Known herpetic keratitis, as determined from history, exam, or microbiological testing
* Known fungal keratitis, as demonstrated from corneal scrapings
* Corneal perforation or impending corneal perforation
* Prior therapeutic keratoplasty for acanthamoeba keratitis
* Unwillingness or inability to follow-up
* No light perception in the affected eye
* Known hypertensive response to steroids
* Corticosteroid allergy
* Concurrent treatment with systemic corticosteroids
* Concurrent granulomatous amoebic encephalitis

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Vision | 6 Months
  Best corrected visual acuity

SECONDARY OUTCOMES:
Self-reported eye pain | 2 months
  Pain scale (Likert 11-point ordinal scale from 0 to 10; 0=no pain, 10=worst pain)
Clinical Resolution | 12 months
  Time until clinical resolution (i.e., healed ocular surface and absence of inflammation)
Multivariate Analysis | 6 Months
  The multivariate analysis will include the following outcomes measured at 6 months: best corrected visual acuity, corneal thinning on optical coherence tomography (OCT), scar density on Scheimpflug imaging, irregular astigmatism, glare, microbial clearance on confocal microscopy, pain score, time until clinical resolution

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Keenan, MD, MPH, Principal Investigator — Proctor Foundation, UCSF; Gerami Seitzman, MD, Principal Investigator — Proctor Foundation, UCSF
Locations (16):
- United States (12):
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington
- Federal University of São Paulo, São Paulo, Brazil
- India (2):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD available on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the main results
Access Criteria: Request by email addressed to principal investigator.